CLINICAL TRIAL: NCT00284193
Title: Combination Therapy of Low Doses of rFVIIa and FEIBA for Severe Hemophilia A Patients With an Inhibitor to Factor VIII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Uriel Martinowitz, Prof. Uri Martinowitz, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3768-UM-CTIL
Record Dates: First submitted 2006-01-17; First posted 2006-01-31 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- feiba-VIIa, hemophilia A-inhibitor therapy (Experimental): COMBINED PATIENT- TAILORED THERAPY WITH CONCOMITANT ADMINISTRATION OF BOTH DRUGS , FOLLOWING EX VIVO THROMBIN GENERATION PREDICTING ASSAYS
  Interventions: Drug: rFVIIa-FEIBA therapy for hemophilia A inhibitors; Drug: FEIBA- Activated Prothrombin Complexes

INTERVENTIONS:
Drug: rFVIIa-FEIBA therapy for hemophilia A inhibitors — DOses tailored per ex vivo spiking thrombin generation
  Other Names: NOVOSEVEN; APCC
Drug: FEIBA- Activated Prothrombin Complexes

SUMMARY:
Patients with severe hemophilia and inhibitors can be treated effectively by Activated Prothrombin Complex Concentrates (APCC, eg. FEIBA) or High dose recombinant factor VIIa (rFVIIa). Rarely, such patients develop refractoriness to these products for whom therapy with sequential FEIBA and rFVIIa has been recently suggested.

The impetus for the present report was a hemophilia A patient with high titer inhibitor (1300BU) who had life threatening hematuria that was resistant to repeated doses of 400µg/kg rFVIIa up to a cumulative dose of 1200 µg/kg given over 6-9 hours.

Thrombin generation (TG) tested in vitro was consistent with resistance to high concentrations of rFVIIa but yielded good response to combinations of low doses of rFVIIa+FEIBA. In a desperate attempt to control the bleeding, concomitant therapy of 25 U/kg FEIBA and 40µg/kg rFVIIa was infused and resulted in arrest of bleeding within minutes. Over a span of about one year the patient has been successfully treated by this combination for more than 200 bleeding episodes in muscles and joints.

DETAILED DESCRIPTION:
Inhibitor patients with HR inhibitors were eligible for study enrollment. After consent blood was drawn and ex- vivo spiked with rFVIIa/FEIBA and combinations, assayed by thrombin generation tests.

The combination yielding sufficient hemostasis was depicted for patients' therapy of future bleeding episodes.

Following actual therapy hemostasis and safety parameters were monitored.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia patients with inhibitors
* Patients signing informed consent

Exclusion Criteria:

* Patients under 16 or above 65
* Patients with allergic reaction or adverse events in previous use the concentrates
* Patients with high risk of thrombosis

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-01; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Hemostasis achieved post therapy | 6-24 hours
  Following acute bleeding therapy hemostasis was defined as good, partial or non-satisfactory
Safety | 0-24 HOURS
  Following therapy presence of any adverse events, especially thromboembolic complications was assessed

SECONDARY OUTCOMES:
Time to Hemostasis | 0-24 HOURS
  Following therapy patients documented time to "GOOD" response

OTHER OUTCOMES:
Coagulation Studies | 0-24 HOURS
  cbc fibrinogen and D-dimer were assessed pre and post therapy, thrombin generation was assayed when possible after 1-2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Uri Martinowitz, MD, Principal Investigator — Sheba Medical Center